CLINICAL TRIAL: NCT04487106
Title: A Phase II Study of Azacitidine, Venetoclax and Trametinib for Patients With Acute Myeloid Leukemia or Higher-Risk Myelodysplastic Syndrome
Brief Title: Azacitidine, Venetoclax, and Trametinib for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia or Higher-Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0506; NCI-2020-05350 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0506 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-21; First posted 2020-07-27 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Chronic Myelomonocytic Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Azacitidine; trametinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Newly Diagnosed AML Patients) (Experimental): INDUCTION (CYCLE 1): Patients receive azacitidine IV over 30-60 minutes or SC on days 1-7, venetoclax PO QD on days 1-28, and trametinib PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION (CYCLES 2-24): Patients receive azacitidine IV over 30-60 minutes or SC on days 1-7, venetoclax PO QD on days 1-21, and trametinib PO QD on days 1-28. Treatment repeats every 28 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Trametinib; Drug: Venetoclax
- Cohort B (Relapsed/Refractory AML or higher-risk MDS or CMML Patients) (Experimental): INDUCTION (CYCLE 1): Patients receive azacitidine IV over 30-60 minutes or SC on days 1-7, venetoclax PO QD on days 1-28, and trametinib PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION (CYCLES 2-24): Patients receive azacitidine IV over 30-60 minutes or SC on days 1-7, venetoclax PO QD on days 1-21, and trametinib PO QD on days 1-28. Treatment repeats every 28 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Trametinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial investigates how well azacitidine, venetoclax, and trametinib work in treating patients with acute myeloid leukemia or higher-risk myelodysplastic syndrome that has come back (relapsed) or has not responded to treatment (refractory). Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax and trametinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. The goal of this study is learn if the combination of azacitidine, venetoclax, and trametinib can help to control acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine overall survival rate at 1 year of the regimen in patients with newly diagnosed acute myeloid leukemia (AML). (Cohort A) II. To determine the complete remission (CR)/complete remission without recovery of counts (CRi) rate of the regimen in patients with relapsed/refractory AML or high-risk myelodysplastic syndrome (MDS). (Cohort B)

SECONDARY OBJECTIVES:

I. To assess other efficacy endpoints (CR rate, minimal residual disease negativity by flow cytometry, relapse-free survival, event-free survival, and overall survival).

II. To assess proportion of patients proceeding to hematopoietic stem cell transplantation (HSCT).

III. To determine the safety of the combination regimen.

EXPLORATORY OBJECTIVES:

I. To evaluate the impact of baseline genomic alterations on response and survival of the combination regimen.

II. To evaluate clonal evolution from diagnosis to relapse.

OUTLINE:

INDUCTION (CYCLE 1): Patients receive azacitidine intravenously (IV) over 30-60 minutes or subcutaneously (SC) on days 1-7, venetoclax orally (PO) once daily (QD) on days 1-28, and trametinib PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION (CYCLES 2-24): Patients receive azacitidine IV over 30-60 minutes or SC on days 1-7, venetoclax PO QD on days 1-21, and trametinib PO QD on days 1-28. Treatment repeats every 28 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * Cohort A (frontline): Newly diagnosed AML
  * Cohort B (relapsed/refractory): Relapsed/refractory AML or relapsed/refractory MDS or chronic myelomonocytic leukemia (CMML) that is intermediate-2 or high-risk by the International Prognostic Scoring System with >= 10% blasts harboring a Ras pathway-activating mutation. Eligible mutations include: activating mutations of KIT, HRAS/NRAS/KRAS, BRAF, CBL or PTPN11 or loss of function mutation of NF1. Other mutations not listed here that are anticipated to activate Ras signaling may be considered for enrollment after discussion with the principal investigator (PI)
* Performance status =< 2 (Eastern Cooperative Oncology Group [ECOG] scale)
* Total serum bilirubin =< 2.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the PI
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 3 x ULN, unless due to the underlying leukemia approved by the PI
* Creatinine clearance >= 30 mL/min
* Ability to swallow
* Signed informed consent

Exclusion Criteria:

* Patients suitable for and willing to receive intensive induction chemotherapy (cohort A only)
* Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of improvement despite antimicrobial treatment)
* Patients with a prior or concurrent malignancy whose natural history or treatment is not anticipated to interfere with the safety or efficacy assessment of the investigational regimen may be included only after discussion with the PI
* Consumed strong inducer of CYP3A or p-glycoprotein within 3 days of study enrollment. Agents include but are not limited to: carbamazepine, phenytoin, rifampin, and St. John's wart
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator. Prior recent treatment with corticosteroids, hydroxyurea and/or cytarabine (given for cytoreduction) permitted
* Pregnant women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception throughout the study period and for at least 6 months after the last dose of study drugs. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control throughout the study period and for at least 4 months after the last dose of study drugs. Lactating women (or those planning to breastfeed) should not breastfeed during treatment of trametinib and for at least 2 months after the last dose of trametinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Short, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Newly Diagnosed AML Patients); Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients): INDUCTION (CYCLE 1): Patients receive azacitidine IV over 30-60 minutes or SC on days 1-7, venetoclax PO QD on days 1-28, and trametinib PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION (CYCLES 2-24): Patients receive azacitidine IV over 30-60 minutes or SC on days 1-7, venetoclax PO QD on days 1-21, and trametinib PO QD on days 1-28. Treatment repeats every 28 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity.
  Azacitidine: Given IV or SC
  Trametinib: Given PO
  Venetoclax: Given PO
Period: Overall Study
Arm/Group | Cohort A (Newly Diagnosed AML Patients) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients)
Started | 5 | 16
Completed | 5 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Newly Diagnosed AML Patients) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients) | Total
Number analyzed (Participants) | 5 | 16 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 7 | 8
  >=65 years | 4 | 9 | 13
Age, Continuous [Median (Full Range); unit: years] | 75 [59 to 78] | 67 [24 to 84] | 69 [24 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 4 | 11 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 13 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 16 | 21

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response
Description: Overall response is defined as the number of participants achieving Complete Remission (CR) or Complete Remission without recovery of counts (CRi) CR is Normalization of the peripheral blood and bone marrow with </= to 5 % blasts with a granulocyte count of 1 x 10^9/L or greater and a platelet count of 100 x 10^9/L and complete resolution of all extramedullary disease. CRi is Peripheral blood and marrow results as for CR, but with incomplete recover of counts (platelets < 100 x 10^9/L or neutrophils < 1 x 10^9/L).
Time Frame: Up to 2.5 years
Population: Of the five participants registered on Cohort A, three were evaluable. Of the sixteen participants registered on Cohort B, thirteen were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Newly Diagnosed AML Patients) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients)
Number analyzed (Participants) | 3 | 13
Participants | 2 | 2

2. Secondary Outcome: Minimal Residual Disease Negativity
Description: Will be assessed by flow cytometry and estimated along with 95% credible intervals.
Time Frame: Up to time of relapse, assessed up to 2.5 years
Population: Of the five participants in Cohort A, three were evaluable for response. Of the 16 participants in Cohort B, 13 were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Newly Diagnosed AML Patients) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients)
Number analyzed (Participants) | 3 | 13
Participants | 1 | 1

3. Secondary Outcome: Relapse-free Survival
Description: Relapse-free survival is the time from documented CR/CRi until relapse or death.
Time Frame: From documented CR/CRi until relapse or death, assessed until study completion
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A (Newly Diagnosed AML Patients) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients)
Number analyzed (Participants) | 3 | 13
Months | 19 [5.6 to 32.3] | NA [31.0 to 34.6] — Within the study's follow-up period, less than half of the patients have experienced relapse, so a median RFS hasn't been statistically determined

4. Secondary Outcome: Event-free Survival
Description: Event-free survival is the time from the first day of treatment until any treatment failure (lack of response within 6 cycles of treatment, relapse, or death).
Time Frame: From the first day of treatment until any treatment failure (lack of response within 6 cycles of treatment, relapse, or death), assessed until study completion
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A (Newly Diagnosed AML Patients) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients)
Number analyzed (Participants) | 3 | 13
Months | 1.8 [0.5 to 36.4] | 2.1 [0.2 to 35.9]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the first day of treatment to time of death from any cause.
Time Frame: From the first day of treatment to time of death from any cause, assessed until study completion
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A (Newly Diagnosed AML Patients) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients)
Number analyzed (Participants) | 3 | 13
Months | 2.5 [0.5 to 36.4] | 2.4 [0.5 to 38.6]

6. Secondary Outcome: Number of Participants Proceeding to Hematopoietic Stem Cell Transplantation
Description: Will be totaled based on the number of participants who continue with hematopoietic stem cell transplantation post treatment.
Time Frame: Up to 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Newly Diagnosed AML Patients) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients)
Number analyzed (Participants) | 3 | 13
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed up to 3.5 years, Adverse Events monitored/assessed up to 2.5 years
Arm/Group | Cohort A (Newly Diagnosed AML Patients) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients)
All-Cause Mortality (participants affected / at risk) | 1/5 | 1/16
Serious Adverse Events (participants affected / at risk) | 2/5 | 4/16
Other Adverse Events (participants affected / at risk) | 3/5 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Newly Diagnosed AML Patients) (N=5) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients) (N=16)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Oral ulcers (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (3) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subdural Hemorrhage (General disorders) | 0 (0) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Newly Diagnosed AML Patients) (N=5) | Cohort B (Relapsed/Refractory AML or Higher-risk MDS or CMML Patients) (N=16)
alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Cardiac-General Other (Cardiac disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1)
Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 12 (12)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema limb (General disorders) | 2 (2) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2) | 10 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Infection-Other (Infections and infestations) | 1 (1) | 1 (1)
Mucositis/stomatitis (Gastrointestinal disorders) | 1 (2) | 5 (5)
Muscle weakness, generalized or specific area (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Pain (General disorders) | 0 (0) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04487106/Prot_SAP_001.pdf
  • Informed Consent Form (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT04487106/ICF_002.pdf